CLINICAL TRIAL: NCT03378869
Title: Perioperative Management and Outcomes of Minimally Invasive Esophagectomy- Experience of a High-volume Tertiary Center in Taiwan
Brief Title: Perioperative Management and Outcomes of Minimally Invasive Esophagectomy
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708054RINB
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: esophagectomy — all the included participants had received esophagectomy, either Ivor Lewis or tri-incision, or more complex procedures.

SUMMARY:
The investigators retrospectively reviewed the data of all patients who had undergone esophagectomy and reconstruction in 2015. Patient characteristics, the surgery performed, method of anesthesia, postoperative hospitalization course, and additional surgical interventions were reviewed and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients received esophageal reconstruction in 2015.

Exclusion Criteria:

* age <18
* not malignancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with esophageal cancer undergoing esophageal reconstruction in 2015.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 day after surgery
  rate of 30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Jung Cheng, MD. PHD, Study Chair — Chief of Department of Anesthesiology, National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No